CLINICAL TRIAL: NCT00400270
Title: A Physical Therapy Treatment for Adults Diagnosed With Asthma in Primary Care: a Randomised Controlled Trial
Brief Title: Breathing and Relaxation Exercises for Asthma: a Randomised Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College London Hospitals (Other)
Collaborators: Welwyn Hatfield Primary Care Trust (Other); University College, London (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC03660
Record Dates: First submitted 2006-11-15; First posted 2006-11-16 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2006-11

CONDITIONS: Asthma
Keywords: Asthma; Randomised controlled trial; Breathing exercises; Relaxation exercises; Primary care
MeSH Terms: conditions — Asthma | interventions — Respiration

INTERVENTIONS:
Procedure: Breathing and relaxation exercises: the Papworth Method

SUMMARY:
All patients on the GP asthma database in one practice were invited for an asthma physical-therapy assessment, at baseline. Volunteers satisfying the inclusion criteria ie - aged between 16 and 70, able to understand, read and write English, give informed consent, willing to attend the surgery to take part in the trial and with no other serious conditions - were invited to participate in the study. Patients were randomised either to a control group, receiving 2 more assessments at 6 and 12 months, or for comparison to a group receiving 5 physical-therapy treatments of integrated breathing and relaxation exercises (known as the Papworth Method (PM)). The two groups would then be compared at 6 and 12 months.

Hypotheses:

1. The PM of breathing and relaxation training would improve the quality of life for adult patients with asthma in primary care, compared with patients only receiving usual medical care.
2. Anxiety and depression, and symptoms from dysfunctional breathing would reduce compared with the control group.
3. Respiratory function measurements would improve compared with the control group.

ELIGIBILITY:
Inclusion Criteria:

* doctor diagnosed asthma, volunteers from the practice asthma database
* 16-70 years of age
* able to understand, speak and write English
* willing to give informed consent
* willing and able to attend the surgery for assessments and treatments

Exclusion Criteria:

* serious co-morbid conditions

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56
Dates: Start 2004-10; Study Completion 2006-01

PRIMARY OUTCOMES:
Health related Quality of Life as measured by the St George's Respiratory Questionnaire

SECONDARY OUTCOMES:
Anxiety and Depression as measured by the Hospital Anxiety and Depression Scale.
Symptoms from dysfunctional breathing measured by the Nijmegen Questionnaire.
Respiratory measurements as measured by spirometry and capnography.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Robert West, PhD, Study Director — Department of Epidemiology and Public Health, University College London
Locations (1):
- Bridge Cottage Surgery, Welwyn, Hertfordshire, United Kingdom